CLINICAL TRIAL: NCT00858000
Title: Analysis of the Incidence of Expression of a Specific Set of Genes and of Tumor Antigens in Cancer Tissue From Patients With Hepatocellular Carcinoma
Brief Title: Analysis of Expression of Specific Markers in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: 111722
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: markers; expression analysis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — This retrospective study is based upon the analysis of archived samples and patient-related data already available at the investigational site

GROUPS / COHORTS (1):
- Group A: No intervention
  Interventions: Other: Retrospective analysis of already archived samples

INTERVENTIONS:
Other: Retrospective analysis of already archived samples — RNA extracted from tissue samples already archived

SUMMARY:
Hepatocellular carcinoma is an aggressive disease with limited therapeutic options. Therefore, new approaches to treat this type of cancer are needed with immunotherapy potentially being one of these. As a first step in the development of novel therapies, expression analysis of specific markers, including tumor antigens will be carried out. This will be done retrospectively using available hepatocellular carcinoma tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* The patient had pathologically proven hepatocellular carcinoma
* All the data required are available from patient's records
* A sufficient amount of RNA is available for all three tissue samples

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
This study will also analyze whether this gene-expression signature is present in matched cirrhotic tissue and the interface tissue with the tumor. | At the time of analysis.
Proportion of hepatocellular carcinoma cancer patients whose tumor tissue -expresses any one or more of specific target antigens -overexpresses c-MET -expresses a pre-defied gene-expression signature | At the time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Florence, Tuscany, Italy